CLINICAL TRIAL: NCT02379793
Title: Skin Irritation Test of LEO 80185 Gel (Calcipotriol Hydrate Plus Betamethasone Dipropionate) in Healthy Japanese Subjects
Brief Title: Skin Irritation Test of LEO 80185 Gel in Healthy Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LP0076-1080
Record Dates: First submitted 2015-02-26; First posted 2015-03-05 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2015-02

CONDITIONS: Skin and Connective Tissue Diseases
Keywords: LEO 80185 gel; calcipotriol; betamethasone
MeSH Terms: conditions — Skin and Connective Tissue Diseases | interventions — Mineral Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LEO 80185 gel, vehicle, liquid paraffin (Experimental): Each subject has all 3 treatments applied topically at the same time. However, the location on which the treatments are applied is randomised in an investigator blinded manner.
  Interventions: Drug: LEO 80185 gel, vehicle, liquid paraffin

INTERVENTIONS:
Drug: LEO 80185 gel, vehicle, liquid paraffin — Each subject has all 3 treatments applied at the same time. Each treatment is applied once to 2 locations on the subject.

SUMMARY:
The purpose of the study is to investigate skin irritation of LEO 80185 gel, gel vehicle and Liquid Paraffin in healthy Japanese male subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent has been obtained.
2. Healthy Japanese male subjects.
3. Aged 20 to 40 years inclusive.
4. Subjects without signs of skin irritation/disease/disorders/symptoms or blemishes on test sites (e.g. erythema, dryness, roughness, scaling, scars, moles, sunburn).
5. Subjects without a significant abnormality, as judged by the (sub)investigator

Exclusion Criteria:

1. Body Mass Index outside the range 18-25 kg/m²
2. History of alcohol or drug abuse.
3. History of allergic reaction to any medications.
4. Any disease that could in any way confound assessment of the test sites.
5. Known or suspected hypersensitivity to any component of LEO 80185 gel.
6. Known or suspected hepatic, renal or cardiac disorders.
7. Known or suspected disorders of calcium metabolism associated with hypercalcaemia or albumin-corrected serum calcium above the reference range from the sample taken during screening.
8. Subjects suspected of infection based on the infection testing results from the sample taken during screening (Hepatitis B surface antigen, HCV antibody, HIV antigen/antibody, serological test for syphilis).
9. Use of systemic, locally injected or inhaled corticosteroids within 4 weeks of Day 1.
10. Use of vitamin D or calcium supplements, or systemic vitamin D analogues within 4 weeks of Day 1.
11. Use of any medication (systemic or topical) within 2 weeks of Day 1.
12. Subjects who have received treatment with any non-marketed drug substance (i.e. an agent which has not yet been made available for clinical use following registration) within 4 weeks or 5 half-lives of Day 1, whichever is longest.
13. Current participation in any other interventional clinical trial.
14. Previously enrolled in this clinical trial.
15. Previous or current photo-induced or photo-aggravated disease (e.g. abnormal response to sunlight).
16. Exposure to excessive or chronic ultraviolet radiation (e.g. sunlight, sun lamps, tanning booths or photo-therapy) within 4 weeks of Day 1.
17. Subjects (or their partner) not using an adequate method of contraception during the trial (Day 1-4).
18. In the opinion of the (sub)investigator, participation in the trial is inappropriate.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2015-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Skin irritation measured as -, +/-, +, ++, +++, ++++ | 4 days

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Co. LTA HAKATA Clinic, Random Square 5F, 6-18 Tenyamachi, Hakata-ku, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en